CLINICAL TRIAL: NCT04448171
Title: Transcutaneous Electric Nerve Stimulation For Pain Control During Office Intra-detrusor Onabotulinumtoxin A Cystoscopy Injection for Overactive Bladder: A Phase III Randomized Controlled Trial
Brief Title: TENS Used for Pain Management During Office Cystoscopy Botox Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Occhino, Associate Professor of Obstetrics and Gynecology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-003510
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Botox injection - bladder; TENS
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the physician administering the Botox, and the study coordinator (outcomes assessor) assigned to the study will be blinded to the randomization. Both groups of participants will receive the TENS unit electrode placement by the assigned clinical nurse who is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Activated TENS Unit with standard pain control measures (Active Comparator): Activated TENS Unit with standard pain control measures during Office Based Cystoscopic Intra-detrusor Onabotulinumtoxin A Injection
  Interventions: Device: Active TENS
- Sham TENS Unit with standard pain control measures (Placebo Comparator): Sham TENS Unit with standard pain control measures during Office Based Cystoscopic Intra-detrusor Onabotulinumtoxin A Injection
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: Active TENS — Standard TENS unit with four pads affixed to the lower back area, will be used in this arm. The TENS device will be set to an active setting.
  Arms: Activated TENS Unit with standard pain control measures
Device: Sham TENS — Standard TENS unit with four pads affixed to the lower back area, will be used in this arm. The TENS device will be set to an inactive setting.
  Arms: Sham TENS Unit with standard pain control measures

SUMMARY:
The purpose of this study is to determine how Transcutaneous Electric Nerve Stimulation (TENS) units affects pain management during office cystoscopic Botox injections and patient satisfaction with the procedure .

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a symptom complex pronounced by urinary urgency, affecting up to 12% of the adult population, with a significant negative impact quality on the life. Cystoscopic intra-detrusor onabotulinumtoxin A is used for the treatment of OAB in participants who do not tolerate or adequately respond to oral anticholinergic medications. The response to the onabotulinumtoxin A injection is transient and requires repeat injections roughly every 6-7 months. Adequate pain control during this procedure is essential for success in the office setting.

Options for adequate pain control during office-based cystoscopy procedures are limited. Currently, varying pain control strategies are being used including local anesthesia (intra-urethral lidocaine, intra-vesicular lidocaine solution), distraction techniques (conversation/music/'squeeze balls'), aromatherapy, intramuscular analgesia, sedation and a combination of these techniques. Despite this, participants often experience pain during the procedure. Trans-cutaneous Electrical Nerve Stimulation (TENS) is a non-pharmacologic, non-invasive and safe method of pain control that involves delivery of electrical impulses to the skin, resulting in a reduction in perceived pain. TENS units have been successfully used for procedural pain management during office hysteroscopy and office colonoscopy. TENS may also help reduce pain during office cystoscopy.

The study is a two arm phase III double-blind, randomized, placebo-controlled trial looking at the effect of TENS unit on pain in participants receiving office based cystoscopic onabotulinum toxin A injection for overactive bladder at the Mayo Clinic in Rochester, Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18 years or older
* Scheduled to receive intra-detrusor Onabotulinumtoxin-A injection for Overactive Bladder in the outpatient clinic
* Reads, speaks, and understands the English language
* Able to understand the requirements of the study, including randomization
* Willing and able to provide written informed consent

Exclusion Criteria:

* Previous use of TENS therapy within one year prior to study enrollment
* Allergy to adhesives
* Currently has an implanted pacemaker or automatic cardiac defibrillator
* History of epilepsy
* Currently pregnant or within 12 weeks postpartum
* Unwilling to be randomized

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Occhino, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were not randomized as they screen failed prior to randomization taking place.
Groups:
- Activated TENS Unit With Standard Pain Control Measures: Activated TENS Unit with standard pain control measures during Office Based Cystoscopic Intra-detrusor Onabotulinumtoxin A Injection
  Active TENS: Standard TENS unit with four pads affixed to the lower back area, were used in this arm. The TENS device was set to an active setting.
- Sham TENS Unit With Standard Pain Control Measures: Sham TENS Unit with standard pain control measures during Office Based Cystoscopic Intra-detrusor Onabotulinumtoxin A Injection
  Sham TENS: Standard TENS unit with four pads affixed to the lower back area, were used in this arm. The TENS device was set to an inactive setting.
Period: Overall Study
Arm/Group | Activated TENS Unit With Standard Pain Control Measures | Sham TENS Unit With Standard Pain Control Measures
Started | 20 | 20
Completed | 18 | 20
Not Completed | 2 | 0
Not completed — Procedure Cancelled | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active TENS: Receive TENS therapy
- Sham TENS: No TENS therapy received
- Total: Total of all reporting groups
Arm/Group | Active TENS | Sham TENS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 72 [49 to 87] | 72 [60 to 84] | 72 [49 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Participant Reported Pain Score From Baseline to Intra-Procedure
Description: Using the participant-reported numerical pain scale, the change in participant reported pain was measured. This change was measured between two time points, baseline and intra-procedure. The participant-reported pain scale ranges from 0 (no pain) to 10 (worst pain) with higher scores indicating worse pain. When analyzing the data, the scale was multiplied by a factor of 10 to get a 100-point scale. Final results are reported using the 100-point scale ranging from 0 (no pain) to 100 (worst pain) with higher scores indicating worse pain.
Time Frame: Baseline; intra-procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activated TENS Unit With Standard Pain Control Measures | Sham TENS Unit With Standard Pain Control Measures
Number analyzed (Participants) | 14 | 17
score on a scale | 27.9 (26.4) | 37.5 (38.2)

2. Secondary Outcome: Change in Participant Satisfaction From Post Procedure to 10 Minutes Following Completion of Cystoscopy
Description: Using the 10-point Likert scale, the change in participant satisfaction was measured. This change was measured between two time points, post procedure and 10 minutes following completion of cystoscopy. Scores on the Likert scale range from 1 (complete dissatisfaction) to 10 (complete satisfaction), with higher scores indicating higher satisfaction.
Time Frame: Postprocedure, 10 minutes following completion of cystoscopy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activated TENS Unit With Standard Pain Control Measures | Sham TENS Unit With Standard Pain Control Measures
Number analyzed (Participants) | 14 | 17
score on a scale | 9.2 (2.0) | 8.5 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 2 weeks.
Arm/Group | Activated TENS Unit With Standard Pain Control Measures | Sham TENS Unit With Standard Pain Control Measures
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Activated TENS Unit With Standard Pain Control Measures (N=20) | Sham TENS Unit With Standard Pain Control Measures (N=20)
Minor Skin Reaction (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04448171/Prot_SAP_000.pdf